CLINICAL TRIAL: NCT00528255
Title: A Multicenter, Open-Label, Phase II Study of the Pharmacokinetics and Safety of the100 Mcg Misoprostol Vaginal Insert (MVI 100) in Women Requiring Cervical Ripening and Induction of Labor
Brief Title: Pharmacokinetics and Safety of the 100 Mcg Misoprostol Vaginal Insert (MVI 100)
Acronym: Miso-Obs-203
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PK portion will be included in a future protocol
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Miso-Obs-203
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Ripening; Induction of Labor
Keywords: cervical ripening; induction of labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Misoprostol Vaginal Insert (MVI 100)

INTERVENTIONS:
Drug: Misoprostol Vaginal Insert (MVI 100) — The MVI 100 is misoprostol 100 mcg, formulated in a sustained release, nonbiodegradeable hydrogel polymer, with a polyester knit retrieval tape; IV oxytocin is permitted ad lib 30 minutes following removal of the MVI assuming no contraindications.
  Other Names: Cervical ripener

SUMMARY:
This study will provide pharmacokinetic data for the MVI 100 (100 mcg) misoprostol vaginal insert when administered to nulliparous women at term gestation requiring cervical ripening and induction of labor.

DETAILED DESCRIPTION:
PK study in women requiring cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at ≥36 weeks 0 days inclusive gestation;
* Aged 18 years or older;
* Candidate for pharmacologic induction of labor;
* Singleton pregnancy;
* Baseline modified Bishop score <4 (see Appendix B);
* Nulliparous (nulliparous is defined as no previous births live or dead after 24 weeks gestation);
* Written informed consent.

Exclusion Criteria:

* Women with hemoglobin level < 11.0 g/dL (confirmed within one week of study drug insertion);
* Women in active labor;
* Presence of uterine or cervical scar or uterine abnormality e.g. bicornate uterus. Biopsies, including cone biopsy of the cervix, are permitted;
* Administration of oxytocin or any cervical ripening or labor inducing agents (including mechanical methods) or a tocolytic drug within 7 days prior to enrollment. Magnesium sulfate is permitted if prescribed as treatment for pre-eclampsia or pregnancy inducted hypertension;
* Severe pre-eclampsia marked by CNS findings, HELLP syndrome, or other end-organ affliction;
* Suspected or confirmed cephalopelvic disproportion and/or fetal malpresentation;
* Diagnosed fetal abnormalities;
* Suspected or confirmed intrauterine growth retardation (less than 10% estimated fetal weight for dates);
* Any evidence of fetal compromise at baseline (e.g., non-reassuring fetal heart rate pattern or meconium staining);
* Receipt of NSAID (including aspirin) within 4 hours of study treatment;
* Ruptured membranes ≥48 hours prior to the start of treatment or suspected chorioamnionitis;
* Fever (oral or aural temperature > 37.5C);
* Any condition in which vaginal delivery is contraindicated e.g., placenta previa or any unexplained genital bleeding at any time after 24 weeks during this pregnancy;
* Known or suspected allergy to misoprostol, dinoprostone, other prostaglandins or any of the excipients;
* Any condition urgently requiring delivery;
* Unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The levels of misoprostol acid in plasma at time points 0 (baseline), 2, 4, 6, 8, 10 and 14 hours. Not all patients will have all in situ time points as the insert may be removed earlier for safety or efficacy reasons. | 24 Hours

SECONDARY OUTCOMES:
-The levels of misoprostol acid in plasma at time of removal, and 30 and 60 minutes post removal. -Assess all adverse events. | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wininger, MD, Principal Investigator — Precision Trials; Arlen Jarrett, MD, Principal Investigator — South Valley Women's Research; Deborah Wing, MD, Principal Investigator — UCI Medical Center/Long Beach Memorial Hospital; Raymond Brown, MD, Principal Investigator — Temple University Hospital; James Byrne, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (6):
- United States (6):
  - Paradise Valley Hospital, Phoenix, Arizona
  - Long Beach Memorial Hospital, Long Beach, California
  - UCI Medical Center, Orange, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Jordan Valley Hospital, West Jordan, Utah